CLINICAL TRIAL: NCT02562378
Title: Phase I Multicenter Clinical Trial Evaluating the Combination of Trastuzumab Emtansine (T-DM1) and Non-pegylated Liposomal Doxorubicin in HER2-positive Metastatic Breast Cancer
Brief Title: T-DM1 and Non-pegylated Liposomal Doxorubicin in Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Breast Cancer
Acronym: THELMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Roche Pharma AG (Industry); Experior (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP038; 2014-001056-28 (EudraCT Number)
Record Dates: First submitted 2015-09-17; First posted 2015-09-29 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): Trastuzumab emtansine (T-DM1) will be administered at a fixed dose of 3.6 mg/kg IV on Day 1 every 3 weeks and three cohorts of patients with three different dose levels of conventional non-pegylated liposomal doxorubicin (45 mg/m2, 50 mg/m2 and 60 mg/m2) IV
  Interventions: Drug: Trastuzumab and non-pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Trastuzumab and non-pegylated liposomal doxorubicin — 3 Cohorts (3+3 design):
  Cohort 1- Trastuzumab 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin (45 mg/m2) IV
  Cohort 2- Trastuzumab 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin (50 mg/m2) IV
  Cohort 3- Trastuzumab 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin (60 mg/m2) IV
  Other Names: T-DM1 and non-pegylated liposomal doxorubicin

SUMMARY:
The primary goal is to determine the maximum tolerated dose (MTD) of the combination of T-DM1 and non-pegylated liposomal doxorubicin in metastatic breast cancer (mBC) patients previously treated with taxanes and trastuzumab-based therapy.

In addition, pharmacokinetic data on the combination of T-DM1 and liposomal doxorubicin will be obtained.

DETAILED DESCRIPTION:
Subjects: Age ≥ 18 years with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer that have relapsed or progressed on or after taxanes and trastuzumab-based therapy. Subjects must have histologic or cytologic confirmation of the HER2-positive metastatic breast cancer. Evidence of measurable or evaluable metastatic disease is required.

Primary objective:

* To determine the maximum tolerated dose (MTD) of the combination of T-DM1 and non-pegylated liposomal doxorubicin in metastatic breast cancer (mBC) patients previously treated with taxanes and trastuzumab-based therapy.

Secondary objectives:

* To determine the efficacy of the combination of T-DM1 and non-pegylated liposomal doxorubicin, defined by the overall response rate (ORR), clinical benefit rate (CBR), number of progressions and number and reasons for deaths.
* To assess the safety profile of the combination of T-DM1 and non-pegylated liposomal doxorubicin, defined by all toxicities reported during the study.
* To evaluate the cardiac safety of the combination of T-DM1 and non-pegylated liposomal doxorubicin measured by left ventricular ejection fraction (LVEF) as assessed by echocardiography, cardiac troponin I and B-type natriuretic peptide (BNP) levels.
* To evaluate the potential role of single nucleotide polymorphisms (SNP) in the predisposition for developing cardiotoxicity.
* To analyze the pharmacokinetics (PK) profile of T-DM1 and its metabolites and non-pegylated liposomal doxorubicin.

Type of study: This is a prospective dose-finding, multicenter and open-label phase I clinical trial.

Treatment: Trastuzumab emtansine (T-DM1) will be administered at a fixed dose of 3.6 mg/kg IV on Day 1 every 3 weeks and three cohorts of patients with three different dose levels of conventional non-pegylated liposomal doxorubicin (45 mg/m2, 50 mg/m2 and 60 mg/m2) IV on Day 1 in cycles of 21 days each are planned.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient able and willing to comply with protocol
* Cytologically or histologically confirmed carcinoma of the breast.
* Incurable locally advanced or metastatic disease who have previously received up to two previous chemotherapy regimens in this setting. Patient must have progressed or relapsed on or after taxane and trastuzumab-based therapy.
* HER2-positive disease
* At least one measurable lesion according to RECIST version 1.1; or patients with non measurable lesions could be included with these exceptions:

  o patients with only blastic bone lesions / with only pleural, peritoneal or cardiac effusion, or meningeal carcinomatosis
* ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Life expectancy ≥ 3 months
* Adequate bone marrow function:

  * Hemoglobin ≥ 10 g/dl.
  * Absolute neutrophil count ≥ 1.5 x 109/L.
  * Platelets ≥ 100 x 109/L without transfusions within 21 days
  * International normalized ratio (INR) < 1.5 × the upper limit of normal (ULN).
* Adequate hepatic and renal function
* Adequate cardiovascular function with LVEF ≥ 55%
* Recovery from all reported toxicities of previous anti-cancer therapies to baseline or grade ≤ 1 (CTCAE version 4.0), except for alopecia
* For women of childbearing potential and not postmenopausal, and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy, and men with partners of childbearing potential, use of forms of contraception

Exclusion Criteria:

* Previous treatment with T-DM1 or anthracyclines
* More than two chemotherapeutic regimens for locally advanced incurable disease or metastatic disease
* Prior anti-cancer treatment with chemotherapy, immunotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin-C), hormonal therapy or lapatinib within 7 days, prior trastuzumab within 21 days (7 days if weekly trastuzumab) or any other targeted therapy within the last 21 days prior to starting study treatment
* Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or mBC is not allowed if:

  * The last fraction of radiotherapy has been administered within 21 days prior to first study drug administration (except for brain irradiation; at least 28 days will be required)
  * More than 25% of marrow-bearing bone has been irradiated
* History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to the active substance or to any of the excipients of T-DM1 or non-pegylated liposomal doxorubicin
* Patients with central nervous system (CNS) involvement. However, patients with metastatic CNS tumors may participate in this trial if the patient is > 4 weeks from radiotherapy completion, is clinically stable with respect to CNS tumor at the time of study entry and is not receiving steroid therapy for brain metastases
* Severe/uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Cardiopulmonary dysfunction
* Current peripheral neuropathy of Grade ≥ 3 per the NCI CTCAE, v4.0
* History of a decrease in LVEF to < 40% or symptomatic congestive heart failure (CHF) with previous trastuzumab treatment
* Prior malignancy, other than carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was cured ≥ 5 years before first dose of study drug with no subsequent evidence of recurrence
* Current known active infection with HIV, hepatitis B, and/or hepatitis C virus
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, MD, Study Director — Hospital Ramon y Cajal, Madrid, Spain
Locations (3):
- MedSIR investigative site, Paris, France
- Spain (2):
  - MedSIR investigative site, Barcelona
  - MedSIR investigative site, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2): Trastuzumab emtansine (T-DM1) will be administered at a fixed dose of 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin at a dose level of 45 mg/m2.
- Period 2: Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2): Trastuzumab emtansine (T-DM1) will be administered at a fixed dose of 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin at a dose level of 50 mg/m2.
- Period 3: Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2): Trastuzumab emtansine (T-DM1) will be administered at a fixed dose of 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin at a dose level of 60 mg/m2.
Period: Overall Study
Arm/Group | Period 1: Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Period 2: Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Period 3: Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Started | 3 | 3 | 9
Completed | 3 | 3 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2): Trastuzumab and non-pegylated liposomal doxorubicin: Trastuzumab 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin (45 mg/m2) IV
- Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2): Trastuzumab and non-pegylated liposomal doxorubicin: Trastuzumab 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin (50 mg/m2) IV
- Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2): Trastuzumab and non-pegylated liposomal doxorubicin: Trastuzumab 3.6 mg/kg IV on Day 1 every 3 weeks and non-pegylated liposomal doxorubicin (60 mg/m2) IV
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2) | Total
Number analyzed (Participants) | 3 | 3 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.5) | 58.7 (2.1) | 45.9 (12.5) | 49.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 9 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 0 | 1 | 2 | 3
  Spain | 3 | 2 | 5 | 10
  Slovenia | 0 | 0 | 2 | 2
ECOG Performance Status (ITT) [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) criteria used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient. ECOG 0 (Fully active) > ECOG 5 (Dead).
  participants
    ECOG score 0 (Fully active) | 3 | 3 | 7 | 13
    ECOG score 1 (Restricted physical activity) | 0 | 0 | 2 | 2
Prior Medication [Count of Participants; unit: Participants] — History of patients treatment that may be concomitant to study treatment, or may limit current treatment.
  Participants
    No | 0 | 0 | 5 | 5
    Yes | 3 | 3 | 4 | 10
Estrogen Receptor (ER) (ITT) [Count of Participants; unit: Participants]
  Positive | 2 | 3 | 6 | 11
  Negative | 1 | 0 | 3 | 4
Progesterone Receptor (PgR) (ITT) [Count of Participants; unit: Participants]
  Positive | 1 | 2 | 4 | 7
  Negative | 2 | 1 | 5 | 8
Human Epidermal Growth Factor Receptor 2 (HER2) (ITT) [Count of Participants; unit: Participants] | 3 | 3 | 9 | 15
HER2 detection method [Count of Participants; unit: Participants]
  Immunohistochemistry (IHC) | 2 | 2 | 7 | 11
  Fluorescence in situ hybridization (FISH) | 1 | 1 | 1 | 3
  Chromogenic in situ hybridization (CISH) | 0 | 0 | 1 | 1
TNM Staging (ITT) [Count of Participants; unit: Participants] — A system to describe the amount and spread of cancer in a patient's body (T= primary tumor size and nature, N= regional lymph node involvement, M= level of metastasis).
  Participants
    Core biopsy | 3 | 3 | 7 | 13
    Fine needle aspiration | 0 | 0 | 1 | 1
    Missing | 0 | 0 | 1 | 1
TNM Staging T Category [Count of Participants; unit: Participants] — T-staging= primary tumor size, location, and nature. Tx means no information, T0= no evidence of tumor. T1-4= Increasing size/location/nature.
  Participants
    Tx | 0 | 0 | 2 | 2
    T1 | 1 | 0 | 3 | 4
    T2 | 0 | 1 | 1 | 2
    T3 | 2 | 1 | 2 | 5
    T4 | 0 | 1 | 1 | 2
TNM Staging N Category [Count of Participants; unit: Participants] — N-staging= spread of tumor into local lymph nodes. Nx means no information, N0= no local involvement. N1-3= Increasing spread into lymph nodes.
  Participants
    Nx | 0 | 0 | 2 | 2
    N0 | 0 | 1 | 1 | 2
    N1 | 0 | 0 | 6 | 6
    N2 | 3 | 2 | 0 | 5
TNM Staging M Category [Count of Participants; unit: Participants] — M-staging= tumor spread to distant organs or tissues. Mx means no information available. M0= No evidence of spread detected, M1= cancer detected in distant organs or tissues.
  Participants
    Mx | 0 | 0 | 2 | 2
    M0 | 0 | 0 | 4 | 4
    M1 | 3 | 3 | 3 | 9
Disease Stage at Initial Diagnostic [Count of Participants; unit: Participants] — Clinical staging is based on information gained up to the initial definitive treatment. Pathologic staging includes clinical information and information obtained from pathologic examination of resected primary and regional lymph nodes. A higher cancer stage, i.e., Stage IV, is more aggressive and typically more difficult to treat.
  Participants
    I | 0 | 0 | 1 | 1
    II | 0 | 0 | 2 | 2
    III | 0 | 0 | 3 | 3
    IV | 3 | 3 | 3 | 9
Metastasis sites (ITT) [Number; unit: participants]
  Metastasis | 3 | 3 | 9 | 15
  Lymph node | 2 | 1 | 7 | 10
  Bone | 3 | 3 | 4 | 10
  Liver | 0 | 2 | 4 | 6
  Lung | 0 | 1 | 4 | 5
  Brain | 1 | 0 | 1 | 2
  Skin | 0 | 0 | 2 | 2
  Other sites | 0 | 1 | 1 | 2
Previous Treatment for Metastatic Breast Cancer [Count of Participants; unit: Participants]
  1 | 0 | 3 | 8 | 11
  2 | 3 | 0 | 0 | 3
  3 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hematological - Dose Limiting Toxicities
Description: Treatment-related adverse events (AEs) of any grade reported in ≥10% of patients.
Time Frame: Baseline up to 6 weeks after patient entry (Cycle2Day21)
Measure: Number; unit: participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
participants
  Neutropenia | 1 | 3 | 7
  Thrombopenia | 1 | 2 | 6
  Anemia | 1 | 1 | 4
  Leukopenia | 0 | 1 | 2
  Lymphopenia | 0 | 1 | 2
  Decreased hemoglobin | 1 | 1 | 0
  Decreased lymphocyte count | 0 | 1 | 1

2. Primary Outcome: Non-Hematological - Dose Limiting Toxicities
Description: Treatment-related AEs of any grade reported in ≥10% of patients.
Time Frame: Baseline up to 6 weeks after patient entry (Cycle2Day21)
Measure: Number; unit: participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
participants
  Asthenia | 3 | 2 | 4
  Nausea | 2 | 3 | 4
  Inc. aspartate aminotransferase | 1 | 1 | 6
  Inc. alanine aminotransferase | 1 | 1 | 4
  Inc. brain natriuretic peptide | 0 | 2 | 4
  Inc. gamma-glutamyl transferasehemoglobin | 2 | 2 | 2
  Increased troponin Ilymphocyte count | 0 | 1 | 4
  Decreased appetite | 1 | 1 | 3
  Alopecia | 0 | 1 | 3
  Epistaxis | 0 | 1 | 2
  Rhinorrhea | 0 | 1 | 2
  Headache | 0 | 2 | 0
  Fatigue | 0 | 0 | 2
  Mucosal inflammation | 0 | 0 | 2
  Inc. blood alkaline phosphatase | 0 | 1 | 1
  Aphthous ulcer | 0 | 1 | 1
  Constipation | 1 | 0 | 1
  Diarrhea | 1 | 0 | 1
  Dry mouth | 0 | 1 | 1
  Gingival bleeding | 0 | 0 | 2
  Vomiting | 0 | 1 | 1
  Hypoalbuminemia | 0 | 1 | 1
  Rash | 0 | 1 | 1

3. Secondary Outcome: Overall Response Rate
Description: Patients with best overall response of confirmed complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST criteria guidelines (version 1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Baseline up to 24 months after patient entry
Population: Best Overall Response (percentage of participants) with confirmed complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST v1.1 criteria guidelines
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
percentage of participants | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 33.3 [7.5 to 70.1]

4. Secondary Outcome: Best Overall Response
Description: Patients with best overall response of confirmed complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST criteria guidelines (version 1.1)
Time Frame: Baseline up to 24 months after patient entry
Population: Best Overall Response, n (%)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
Participants
  Partial response | 1 | 2 | 3
  Stable disease ≥24 weeks | 1 | 0 | 3
  Stable disease <24 weeks | 0 | 1 | 2
  Progressive disease | 1 | 0 | 0
  Not evaluable | 0 | 0 | 1

5. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) lasting more than 24 weeks based on local investigator's assessment
Time Frame: Baseline up to 24 months after patient entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
percentage of participants | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 66.7 [38.4 to 88.2]

6. Secondary Outcome: Progression-free Survival
Description: Patients with progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Baseline up to 24 months after patient entry
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
months | 8.2 [1.3 to 10.3] | 7.0 [3.8 to 10.2] | 7.2 [4.5 to 9.6]

7. Secondary Outcome: Grade 3/4 Adverse Events, SAEs, Deaths and Discontinuations
Description: Patients with grade 3/4 adverse events, Serious Adverse Events (SAEs), deaths and discontinuations
Time Frame: Baseline up to 24 months after patient entry
Measure: Number; unit: participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
participants
  Neutropenia | 0 | 2 | 6
  Thrombopenia | 0 | 0 | 2
  Leukopenia | 0 | 1 | 1
  Lymphopenia | 0 | 1 | 1
  Increase in aspartate aminotransferase (AST) | 0 | 0 | 2
  Fatigue | 0 | 0 | 1

8. Secondary Outcome: Discontinuation of the Study Drugs Due to Any Cardiotoxicity
Description: Rate of patients who discontinued treatment due to Cardiac Function or Due to Cardiac Cause
Time Frame: Baseline up to 24 months after patient entry
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 0 | 0

9. Secondary Outcome: Left Ventricular Dysfunction Class IV
Description: New York Heart Association grading of Level II cardiotoxicities characterized by dose-independent reversible myocardial damage.
  The classes used in this system, I to IV with I indicating less severity and higher numbers indicating greater severity.
Time Frame: Baseline up to 24 months after patient entry
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
Participants | 0 | 1 | 2

10. Secondary Outcome: Serum HER-2 Levels
Description: Serum human epidermal growth factor receptor 2 (HER-2) Levels (ng/mL) - Cycle 1 Day 1 and Cycle 4 Day 1.
Time Frame: Baseline and after 4 cycles of treatment (Cycle4Day21)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
ng/mL
  Baseline, Serum HER-2 (ng/mL) | 12.7 (5.8) | 38.1 (35.7) | 17.5 (6.0)
  Cycle 4 Day 21, Serum HER-2 (ng/mL) | 7.4 (0) | 15.2 (0.6) | 18.8 (5.4)

11. Secondary Outcome: Doxorubicinol - Concentration (Cmax)
Description: Plasma concentration of Doxorubicinol using a validated liquid chromatography electrospray tandem mass spectrometry (LC-MS/MS) method
Time Frame: Baseline (Cycle1Day1) and end of Cycle 2 (C2D21)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
μg/mL
  Cycle 1 Day 1 | 14.8 (8.4) | 9.19 (42.1) | 15.2 (70.6)
  Cycle 2 Day 21 | 16.0 (25.2) | 10.1 (38.9) | 15.6 (54.5)

12. Secondary Outcome: Doxorubicinol - Area Under Curve (AUC)
Description: Area under the plasma concentration versus time curve for the pharmacokinetic parameters for doxorubicinol by treatment dose level
Time Frame: Baseline (Cycle1Day1) and end of Cycle 2 (C2D21)
Measure: Mean (Standard Deviation); unit: ng x h/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
ng x h/mL
  Cycle 1 Day 1- AUC | 982 (28.4) | 888 (27.8) | 1340 (65.0)
  Cycle 2 Day 21- AUC | 899 (40.7) | 763 (25.4) | 1100 (50.3)

13. Secondary Outcome: Doxorubicinol - Apparent Half-life (t1/2)
Description: Apparent half-life for doxorubicinol by treatment dose level.
Time Frame: Baseline (Cycle1Day1) and end of Cycle 2 (C2D21)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
days
  Cycle 1 Day 1 | 93.4 (37.9) | 78.5 (6.0) | 69.3 (11.7)
  Cycle 2 Day 21 | 51.91 (0.5) | 64.01 (23.6) | 49.41 (1.9)

14. Secondary Outcome: Doxorubicinol - Tmax
Description: Maximum concentration of drug in plasma (Tmax)
Time Frame: Baseline (Cycle1Day1) and end of Cycle 2 (C2D21)
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
hours
  Cycle 1 Day 1- Tmax | 3.75 [3.58 to 3.75] | 3.58 [3.58 to 3.92] | 3.63 [3.5 to 3.83]
  Cycle 2 Day 21- Tmax | 4.02 [4.00 to 4.23] | 3.58 [1.17 to 4.15] | 3.78 [3.75 to 4.00]

15. Secondary Outcome: Trastuzumab - Cmax
Description: Pharmacokinetic parameters for trastuzumab
Time Frame: Baseline (Cycle1 Day1)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
μg/mL | 94.6 (16.8) | 114 (2.8) | 78.3 (7.6)

16. Secondary Outcome: Trastuzumab - AUC
Description: Pharmacokinetic parameters for trastuzumab
Time Frame: Baseline (Cycle1Day1)
Measure: Mean (Standard Deviation); unit: μg x h/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
μg x h/mL | 348 (14.4) | 372 (30.3) | 317 (18.9)

17. Secondary Outcome: Trastuzumab - Tmax
Description: Pharmacokinetic parameters for trastuzumab
Time Frame: Baseline (Cycle1Day1)
Measure: Mean (Full Range); unit: hours
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
hours | 1.95 [1.83 to 2.00] | 1.83 [1.83 to 2.02] | 1.95 [1.8 to 2.08]

18. Secondary Outcome: DM-1 - Cmax
Description: Pharmacokinetic parameters for emtansine (DM1) by treatment dose level
Time Frame: Baseline (Cycle1Day1)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
μg/mL | 3.76 (18.2) | 8.03 (67.3) | 5.13 (59.1)

19. Secondary Outcome: DM-1 - AUC
Description: Pharmacokinetic parameters for DM1 by treatment dose level
Time Frame: Baseline (Cycle1Day1)
Measure: Mean (Standard Deviation); unit: μg x h/mL
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
μg x h/mL | 23.1 (143.1) | 10.1 (25.0) | 5.63 (24.9)

20. Secondary Outcome: DM-1 - Tmax
Description: Pharmacokinetic parameters for DM1 by treatment dose level
Time Frame: Baseline (Cycle1Day1)
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
Number analyzed (Participants) | 3 | 3 | 9
hours | 2.0 [1.95 to 581] | 1.83 [1.83 to 2.02] | 1.95 [1.80 to 2.08]

ADVERSE EVENTS:
Time Frame: Baseline up to 24 months after patient entry
Arm/Group | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) (N=3) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) (N=3) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2) (N=9)
Infections and infestations (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Appendicitis
Investigations (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Aspartate aminotransferase increased
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Nervous system disorder
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Partial seizures
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Trastuzumab + Doxorubicin (45 mg/m2) (N=3) | Cohort 2, Trastuzumab + Doxorubicin (50 mg/m2) (N=3) | Cohort 3, Trastuzumab + Doxorubicin (60 mg/m2) (N=9)
Asthenia (General disorders) | 3 (3) | 2 (2) | 7 (7) — Weakness or lack of energy.
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) — Walking abnormally compared to usual.
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 7 (7)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 6 (6)
Aspartate aminotransferase (AST) increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 6 (6)
Alanine aminotransferase (ALT) increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4)
Brain natriuretic peptide increased (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4)
Gamma-glutamyltransferase increased (Hepatobiliary disorders) | 2 (2) | 2 (2) | 2 (2)
Troponin increased (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4)
White blood cell count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) — Can also be caused by bile duct obstruction, gallbladder disease, or bone disorders
Haemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Blood albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count abnormal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (5)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (5)
Eye disorders (Eye disorders) | 0 (0) | 1 (1) | 3 (3)
Nervous system disorders (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) — Lack of adequate healthy red blood cells
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) — Sensory pain in any region of the head

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT02562378/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT02562378/SAP_001.pdf